CLINICAL TRIAL: NCT03219606
Title: Impact of Education and Training of Modified Rodnan Skin Scoring on the Reliability of Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Bong Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1715-133-856
Record Dates: First submitted 2017-06-28; First posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Scleroderma, Systemic
Keywords: Systemic sclerosis; Education; Modified Rodnan skin score
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- education arm (Experimental): Participants in education arm will have an organized education course of modified Rodnan Skin Scoring.
  Interventions: Other: Organized education course of Modified Rodnan Skin Scoring

INTERVENTIONS:
Other: Organized education course of Modified Rodnan Skin Scoring — 1. Lecture: An expert rheumatologist (master instructor) give a lecture to explain the technique of Modified Rodnan Skin Scoring (MRSS).
  2. Demonstration: Master instructor demonstrate the patient assessment without revealing his score.
  3. Practical training: Participants assess the MRSS of 8 patients with systemic sclerosis. Two other expert rheumatologists assist the course.

SUMMARY:
The aim of the study is evaluating the efficacy of organized education process of the modified Rodnan Skin Score (MRSS) in the systemic sclerosis. Ten physician in South Korea will be voluntarily enrolled and receive the organized training program, which encompass the lecture and demonstration of skin scoring by expert rheumatologist. Reliability and accuracy of the skin scoring before and after the education will be compared.

DETAILED DESCRIPTION:
1. Participants Ten physicians who are voluntarily enrolled in the organized education course

2. Organized education course

1. Lecture: A expert rheumatologist (master instructor) give a lecture to explain the technique of MRSS.
2. Demonstration: Master instructor demonstrate the patient assessment without revealing his score.
3. Practical training: Participants assess the MRSS of 8 patients with systemic sclerosis. Two other expert rheumatologists

3. Protocol

1. Instructor pre-meeting: Three instructors including master instructor assess the MRSS of 8 systemic sclerosis patients. Modified Rodnan score drawn by arrangement among them is defined as standard score of each patient.
2. Pre-education scoring: Participants assess the MRSS of 8 patients before the education course.
3. Organized education course
4. Post-education scoring: Participants assess the MRSS of the same 8 patients after i) lecture and ii) demonstration of master instructor
5. written test: Participants take written examination regarding the MRSS before and after the education.

4. Outcomes

1. Inter-observer reliability of MRSS before and after the education
2. Change in difference between score measure by each participant and standard score after the educational course.
3. Change in the score of written test after the educational course.

ELIGIBILITY:
Inclusion Criteria:

* Physician who voluntarily enroll the educational program.

Exclusion Criteria:

* Non-physician

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-10-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in difference between score measured by each participant and standard score after the organized education course. | 1. One day before the education course 2. After 20 minutes of the lecture 3. After 20 minutes of the demonstration and practical training

SECONDARY OUTCOMES:
Change in written test score of each participant after the organized education course | 1. One day before the education course 2. After 20 minutes of the lecture 3. After 20 minutes of the demonstration and practical training
Change in inter-observer reliability of MRSS after the organized education course | 1. One day before the education course 2. After 20 minutes of the lecture 3. After 20 minutes of the demonstration and practical training

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Khanna D, Furst DE, Clements PJ, Allanore Y, Baron M, Czirjak L, Distler O, Foeldvari I, Kuwana M, Matucci-Cerinic M, Mayes M, Medsger T Jr, Merkel PA, Pope JE, Seibold JR, Steen V, Stevens W, Denton CP. Standardization of the modified Rodnan skin score for use in clinical trials of systemic sclerosis. J Scleroderma Relat Disord. 2017 Jan-Apr;2(1):11-18. doi: 10.5301/jsrd.5000231. PMID 28516167
- [Result] Czirjak L, Nagy Z, Aringer M, Riemekasten G, Matucci-Cerinic M, Furst DE; EUSTAR. The EUSTAR model for teaching and implementing the modified Rodnan skin score in systemic sclerosis. Ann Rheum Dis. 2007 Jul;66(7):966-9. doi: 10.1136/ard.2006.066530. Epub 2007 Jan 18. PMID 17234649